CLINICAL TRIAL: NCT07187778
Title: Phase II Trial of Single Agent Belzutifan or Pembrolizumab Versus Combination as Neoadjuvant Therapy in Clear Cell Renal Cell Carcinoma (BLAZE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1884; NCI-2025-06635 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combo-B+P: Phase II Combo Neoadjuvant Treatment with Belzutifan (PO/QD) and Pembrolizumab (IV Q3W) (Experimental): Participants will undergo evaluations at baseline, 3 weeks, 6 weeks, 9 weeks, and 12 weeks after initiation of treatment
  Interventions: Drug: Pembrolizumab; Drug: Belzutifan
- Mono-B: Phase II Mono Neoadjuvant Treatment with Belzutifan (PO/QD) (Experimental): Participants will undergo evaluations at baseline, 3 weeks, 6 weeks, 9 weeks, and 12 weeks after initiation of treatment
  Interventions: Drug: Belzutifan
- Mono-P: Phase II Mono Neoadjuvant Treatment with Pembrolizumab (IV Q3W) (Experimental): Participants will undergo evaluations at baseline, 3 weeks, 6 weeks, 9 weeks, and 12 weeks after initiation of treatment
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Oral administration
  Other Names: Keytruda
  Arms: Combo-B+P: Phase II Combo Neoadjuvant Treatment with Belzutifan (PO/QD) and Pembrolizumab (IV Q3W); Mono-P: Phase II Mono Neoadjuvant Treatment with Pembrolizumab (IV Q3W)
Drug: Belzutifan — Oral administration
  Other Names: Welireg
  Arms: Combo-B+P: Phase II Combo Neoadjuvant Treatment with Belzutifan (PO/QD) and Pembrolizumab (IV Q3W); Mono-B: Phase II Mono Neoadjuvant Treatment with Belzutifan (PO/QD)

SUMMARY:
To learn if belzutifan alone, pembrolizumab alone, or belzutifan and pembrolizumab in combination given before a total or partial nephrectomy (surgery to remove all or part of a kidney) can help to control locally advanced ccRCC.

DETAILED DESCRIPTION:
Primary Objective:

1. A composite primary endpoint of objective response rate (ORR) or pathologic response rate (PRR) at 12 weeks after neoadjuvant therapy. objective response - defined as partial [≥ 30% decrease in largest diameter] or complete response on imaging at 12 weeks after neoadjuvant therapy (according to Response Evaluation Criteria In Solid Tumors [RECIST] criteria) (Appendix 14.2)

Pathologic response - defined as ≤25% residual viable tumor in post-therapy pathology specimen.

Secondary Objectives:

1. Relapse-Free Survival (RFS) - defined as the length of time after randomization to date of radiographic/clinical progression, recurrence or death
2. Safety/Tolerability - including adverse events [by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE)], laboratory results, vital signs, physical examinations
3. Quality of Life - as measured by patient-reported outcome measures, including EORTC-QLQ-C30 and FACT-G Single Item GP5 (Appendix 14.3, Appendix 14.4)

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven clear cell renal cell carcinoma (ccRCC).

  a. Extra tissue should be submitted if available for correlative analysis. Formalin-fixed paraffinembedded (FFPE) tissue blocks are preferred to slides. Details pertaining to tumor tissue submission can be found in the Lab Procedures Manual.
* Has intermediate-high risk, high risk, or M1 ccRCC as defined by the following pathological tumor-node metastasis and tumor grading:

Intermediate-high risk ccRCC*

1. pT2 (by radiographic/size criteria), Grade 4 or with sarcomatoid/rhabdoid features (on biopsy), N0, M0
2. pT3 (presence of tumor thrombus, perinephric and/or sinus fat invastion by imaging), any grade, N0, M0 High-risk ccRCC*
3. pT4, any g.rade, N0, M0
4. pT, any stage, any grade, N+, M0 M1 RCC participants who present with the primary kidney tumor, but also solid, isolated, soft tissue metastases that are planned to be completely resected at the time of nephrectomy are eligible (e.g. metastasis to ipsilateral adrenal gland).

   * NOTE: Fuhrman Tumor Grade and/or WHO/ISUP Tumor Grade are required for all subjects entering the study.

     • Evaluated by urology and approved as candidates for nephrectomy.

     • Age ≥18 years and consent to participation.

     • Performance status of 0-1 per Zubrod/Eastern Cooperative Oncology Group [ECOG] scale.

     • Absence of distant metastases on imaging of chest, abdomen and pelvis within 42 days of enrollment (by CT, MRI, or PET imaging). Brain imaging is not required unless clinical suspicion per the treating provider.

     • Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

     • Screening laboratory criteria include the following: a. ANC ≥1000, PLT ≥ 75, Hgb ≥9 (transfusion allowed if Hgb < 1.5 or = to upper limit of normal

     • Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

     • Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (see below) prior to study entry and for the duration of study participation, including for 120 days after the last dose of pembrolizumab and 30 days after the last dose of belzutifan. WOCBP will be required to have a negative pregnancy test prior to cycle 1 day 1 of treatment, ≤24 hours prior to first dose of treatment. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

     • Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 30 days after the last dose of study intervention. The investigator should evaluate the potential for contraceptive method failure (ie, noncompliance, recently initiated) in relationship to the first dose of study intervention. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

     • This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

     o Postmenopausal (no menses in greater than or equal to 12 consecutive months).
     * History of hysterectomy or bilateral salpingo-oophorectomy.
     * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
     * History of bilateral tubal ligation or another surgical sterilization procedure.

       • Male participants are eligible to participate if they agree to the following during the intervention period and for at least 7 days after the last dose of study intervention:

       • Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR

       • Must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause) as detailed below:

       - Agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a WOCBP who is not currently pregnant

   Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.

   - Male participants must also agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person of any sex.

   • Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   • Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of pembrolizumab and 30 days after last belzutifan administration.
   * Ability to understand and the willingness to sign a written informed consent document.

   Exclusion Criteria:
   * Has any of the following:

<!-- -->

1. A pulse oximeter reading <92% at rest, or
2. Requires intermittent supplemental oxygen, or
3. Requires chronic supplemental oxygen

   • Patients who have had chemotherapy or radiotherapy for RCC prior to study.

   • Patients who are receiving any other investigational agents.

   • History of allergic reactions attributed to compounds of similar chemical or biologic composition to belzutifan, pembrolizumab, or other agents used in study.

   • Prior systemic therapy with anti-PD1, PD-L1, PD-L2, or CTLA-4 or received colony-stimulating factors (eg, G-CSF, GM-CSF or recombinant EPO) ≤28 days prior to the first dose of study intervention.
   * Diagnosis of immunodeficiency, active autoimmune disease (per Investigator's discretion), history of pneumonitis, active infection, or known additional malignancy other than RCC.
   * Has a known history of HIV infection. Note: Testing for HIV at screening is only required if mandated by local health authority.
   * Has a known history of HBV (defined as HBsAg reactive) or known active HCV (defined as HCV RNA [qualitative] is detected) infection.

Note: Testing for HBV and HCV is only required if mandated by local health authority.

• Patients who cannot fulfill study requirements for any reason.

* Pregnant or breastfeeding women are excluded from this study because pembrolizumab is a Class-D agent with the potential for teratogenic or abortifacient effects and belzutifan has shown embryofetal toxicity in nonclinical studies
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

  a. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are NOT excluded. Invasive cancers are allowed if treated and in complete remission for at least 3 years.
* Has any known metastatic disease that is not planned to undergo surgical resection at the time of surgery (with the exception of ipsilateral adrenal metastases that are resectable at surgery).
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction ≤6 months from Day 1 of study drug administration, or New York Heart Association Class III or IV congestive heart failure. Medically controlled arrhythmia stable on medication is permitted.
* Has moderate to severe hepatic impairment (Child-Pugh B or C).
* Is unable to swallow orally administered medication or has a gastrointestinal disorder affecting absorption (eg, gastrectomy, partial bowel obstruction, malabsorption).
* Has received prior treatment with belzutifan or another HIF-2α inhibitor.
* Is currently receiving either strong (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate (eg, bosentan, efavirenz, modafinil) inducers of CYP3A4 that cannot be discontinued for the duration of the study.

Note: A current list of strong/moderate inducers of CYP3A4 can be found at the following website:

https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-druginteractionstable-substrates-inhibitors-and-inducers • Has an active infection requiring systemic therapy.

• Has active TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-07-19 (Estimated); Study Completion 2029-07-19 (Estimated)

PRIMARY OUTCOMES:
1. Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org